CLINICAL TRIAL: NCT04117880
Title: Nonsense Mutation Aniridia: An Ataluren (PTC124) Phase 2 Extension Study
Brief Title: A Phase 2 Open Label Extension Study in Participants With Nonsense Mutation Aniridia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study cancelled before protocol was implemented.
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-028e- ANI
Record Dates: First submitted 2019-09-19; First posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-09

CONDITIONS: Aniridia
MeSH Terms: conditions — Aniridia | interventions — ataluren

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ataluren (Experimental): Ataluren Oral suspension taken 3 times per day (10 mg/kg in the morning, 10 mg/kg at mid-day, and 20 mg/kg in the evening).
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — Oral
  Other Names: PTC124

SUMMARY:
This is a Phase 2, multicenter, open-label study evaluating the overall systemic and ocular safety profile of ataluren in nonsense mutation aniridia as determined by the incidences of treatment-emergent adverse events (TEAEs) as well as abnormal findings on laboratory assessments, vital signs, physical examinations, ophthalmoscopy, and slit-lamp examination.

Participants who complete PTC124-GD-028 ANI (NCT02647359) meet all inclusion and none of the exclusion criteria will be enrolled into this study.

DETAILED DESCRIPTION:
This study was a planned extension study of PTC124-GD-028 ANI (NCT02647359) and was never initiated.

ELIGIBILITY:
Inclusion Criteria

Participants who will be selected for this study must meet the following criteria:

1. Evidence of signed and dated informed consent document(s) indicating that the study candidate (and/or a parent/legal guardian) has been informed of all pertinent aspects of the study. Note: If the study candidate is considered a child under local regulation, a parent or legal guardian must provide written consent prior to initiation of study screening procedures and the study candidate may be required to provide written assent. The rules of the responsible institutional review board/independent ethics committee (IRB/IEC) regarding whether one or both parents must provide consent and the appropriate ages for obtaining consent and assent from the participant should be followed.
2. Must have participated in and exited from Study PTC124-GD-028 ANI
3. Age ≥2 years and of either gender.
4. Body weight ≥12 kg.
5. Willingness and ability to comply with scheduled visits, drug administration plan, study procedures, and study restrictions.
6. Good general health.
7. Female participants of childbearing potential are eligible for the study but must be willing to use adequate (at least 1 form of) contraceptive methods as described below during the study treatment period (starting from the day of first dose of study drug and ending 60 days after the last dose of study drug). Childbearing potential is defined as participants who have experienced menarche and who are neither postmenopausal or have been permanently sterilized.

   * Hormonal methods of contraception (including oral and transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing intrauterine contraceptive devices [IUDs]) initiated at least 14 days prior to the first dose of study drug
   * Abstinence
   * Placement of a copper-containing IUD
   * Condom with spermicidal foam/gel/film/cream/suppository
   * Postmenopausal at least 12 months prior to first dose of study drug or permanently sterilized (for example, tubal occlusion, hysterectomy, bilateral salpingectomy)
   * Male partner who has had a vasectomy for at least 3 months prior to the first dose of study drug
8. Male participants with partners of childbearing potential must agree to use the following adequate (at least 1 form of) contraception during the study treatment period (starting from the day of first dose of study drug and ending 60 days after the last dose of study drug):

   * Abstinence
   * Vasectomy for at least 3 months prior to first dose of study drug or surgically sterile
   * Without a vasectomy, must use a condom with spermicidal foam/gel/film/cream suppository

Exclusion Criteria

The presence of any of the following conditions will exclude a participant from study enrollment:

General exclusion criteria

1. Participation in any drug or device clinical investigation (other than Study PTC124-GD-028 ANI) within 90 days prior to Visit 1 (Screening) or anticipation of participating in any other drug or device clinical investigation during this study.
2. Surgery within 30 days prior to enrollment.
3. Female participants who are pregnant or breastfeeding. Female participants of childbearing potential must have a negative pregnancy test (beta-human chorionic gonadotropin [β-HCG]) at screening and must use adequate (at least 1 form of) contraceptive methods.
4. Active ocular infection or inflammation.
5. Prior or ongoing medical condition (for example, concomitant illness, alcoholism, drug abuse, psychiatric condition), medical history, physical findings, or laboratory abnormality that, in the Investigator's opinion, could adversely affect the safety of the participant, makes it unlikely that the course of study drug administration or follow-up would be completed, or could impair the assessment of study results.
6. Participants with a positive result for hepatitis B, hepatitis C, or human immunodeficiency virus at Visit 1 (Screening).

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-31 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | 104 weeks

SECONDARY OUTCOMES:
Change From Baseline in Visual Acuity at Week 104 | 104 weeks
Change From Baseline in Severity of Corneal Keratopathy at Week 104 | 104 weeks